CLINICAL TRIAL: NCT00869648
Title: Head Positions to Open the Upper Airway- a Pilot Study
Brief Title: Head Positions to Open the Upper Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Peter Paal, PD MD MBA EDAIC EDIC, PD MD MBA EDAIC EDIC, Medical University Innsbruck
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UN3371
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Apnea; Cardiopulmonary Resuscitation
Keywords: Airway; Anaesthesia; Resuscitation; Ventilation
MeSH Terms: conditions — Apnea; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neutralposition (Active Comparator): Head placed in neutral position
  Interventions: Procedure: Neutral head position
- Extension (Active Comparator): Head placed in extension
  Interventions: Procedure: Extension
- Anaesthesiologist's position (Active Comparator): Head placed in position deemed optimal by an anaesthesiologist
  Interventions: Procedure: Anaesthesiologist's position

INTERVENTIONS:
Procedure: Extension — After anaesthesia induction the head is placed in extension
  Arms: Extension
Procedure: Neutral head position — After anaesthesia induction the head is placed in neutral position
  Arms: Neutralposition
Procedure: Anaesthesiologist's position — after anaesthesia induction the head is placed in a position deemed optimal by the anaesthesiologist
  Arms: Anaesthesiologist's position

SUMMARY:
Ventilation during basic life support improves survival in cardiac arrest patients significantly. Unfortunately, this is in contrast to the willingness of potential rescuers to perform mouth-to-mouth ventilation. For example, although healthcare professionals would perform mouth-to-mouth ventilation on a 4-year old drowned child in >90% of cases, this likelihood would decrease to ~10% in the case of a young male unconscious patient in a San Francisco public bus. Possibly, lay rescuers would perform assisted ventilation more often if a simple ventilation device were available. However, both the willingness to perform assisted ventilation plus the ability to open and to maintain the airway patent are necessary to ensure efficient ventilation in an unconscious patient with an unprotected upper airway.

Since retention of skills after basic life support classes are notoriously low, a resuscitation tool should incorporate self-explanatory features to improve applicability, and to provide built-in safety. Thus, an option could be to ensure an open airway by the use of a built-in indicator within a ventilating device to confirm correct head extension. One possible approach may be to determine head position angles that make an open airway likely, and integrate these angles into a scale on a ventilating device; however, safe head extension needs to be determined first to prevent harm.

The purpose of this study is to determine head position angles and ventilation parameters reflecting neutral position, maximal extension and a position deemed optimal by an anaesthesiologist in patients undergoing anaesthesia induction for elective surgery in a first step to design a ventilating device to optimise ventilation of an unprotected upper airway. The investigators will ventilate 30 patients with a pillow under the head simulating ventilation in the operating theater, and 30 patients without a pillow under the head simulating ventilation during cardiopulmonary resuscitation.

Dentures will not be removed during assessment. After anaesthesia induction the head will be consecutively flexed in the three positions and measurements performed. Afterwards, general anaesthesia and surgery will ensue. The health risk for this extra minutes of mask ventilation is minimal.

The null hypothesis is that there will be no differences in head position angles and ventilation parameters.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II

Exclusion Criteria:

* Cervical spine pathologies
* Peripheral nerve deficiencies
* Body mass index >40kg/m2
* Obvious primary or secondary craniofacial abnormalities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Head position angles | Within 5 minutes after anaesthesia induction

SECONDARY OUTCOMES:
Tidal volume | Within 5 minutes after anaesthesia induction

CONTACTS AND LOCATIONS:
Overall Officials: Peter Paal, MD, DESA, Principal Investigator — Medical University Innsbruck

REFERENCES:
- [Derived] Mitterlechner T, Paal P, Kuehnelt-Leddhin L, Strasak AM, Putz G, Gravenstein N, von Goedecke A, Wenzel V. Head position angles to open the upper airway differ less with the head positioned on a support. Am J Emerg Med. 2013 Jan;31(1):80-5. doi: 10.1016/j.ajem.2012.06.007. Epub 2012 Sep 1. PMID 22944550